CLINICAL TRIAL: NCT00742911
Title: Phase I Study of Disulfiram and Copper Gluconate for the Treatment of Refractory Solid Tumors Involving the Liver
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI26679
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Cancer
Keywords: Solid Tumors, Liver
MeSH Terms: conditions — Neoplasms | interventions — Disulfiram; Gluconates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Disulfiram; Drug: Copper Gluconate

INTERVENTIONS:
Drug: Disulfiram — Patients will take a pill of disulfiram at a fixed dose of 250 mg with their evening meal. This dose of disulfiram used to treat alcoholism. We will start by administering 2 mg of copper as copper gluconate along with 250 mg disulfiram.
  Patients must not consume beverages containing alcohol while taking disulfiram.
  Other Names: Chemical Name: tetraethylthiuram disulfide; Other names: Antabuse
Drug: Copper Gluconate — Commercially available. Copper gluconate has long been manufactured and sold as a food supplement. Copper gluconate should be taken separately from disulfiram, and if possible with breakfast.
  Copper gluconate should not be administered to individuals with Wilson's disease or a family history of Wilson's disease.
  Patients will receive 2 mg, 4mg, 6mg or 8mg daily
  Other Names: Chemical Name: copper gluconate; Other names: none

SUMMARY:
OBJECTIVES:

Primary Objectives

• Determine the safety and toxicity profile of co-administration of disulfiram and copper gluconate for the treatment of refractory malignancies that have metastasized to the liver.

Secondary Objectives

* Determine if disulfiram and copper gluconate induce measurable responses for the treatment of hepatic metastases from solid tumors.
* Qualitative assessment of the induction of S-glutathionylation in proteins of circulating leukocytes in patients treated with disulfiram and copper gluconate.

DETAILED DESCRIPTION:
We have performed experimental studies demonstrating the anti-cancer efficacy of an old alcoholism treatment drug, disulfiram, combined with supplementation with certain metal ions. Together, disulfiram and metal ions induce S-glutathionylation of critical cancer cell proteins, inhibiting their activity, reducing tumor growth and inducing tumor cell apoptosis. The most active metal ion that can be paired with disulfiram appears to be the divalent metal ion copper. The purpose of this study is to determine the safety of co-administrating the thiocarbamate molecule disulfiram together with copper gluconate to patients with stage IV cancer metastatic to the liver.

Other investigators have studied the effect of disulfiram alone administered to patients with metastatic melanoma, and have observed no clinical benefit when disulfiram is administered without metal ion supplements (Dr. Patrick J. Farmer, University of California Irvine, personal communication).

We therefore propose that the optimum approach to using disulfiram as an antineoplastic agent is to co-administer it with metal ion supplements. While a number of metal ions can enhance the antineoplastic activity of disulfiram, including Zn2+, we have found Cu2+ to be the most active. This observation has been confirmed by others, who have shown that Cu2+ supplementation of growth media increases the pro-apoptotic (Cen 2004) and proteosomal-inhibitory (Chen 2006) activities of disulfiram. Compared to surrounding normal tissue, many cancer cells contain highly elevated levels of copper (Habib 1980; Rizk 1984; Turecky 1984; Diez 1989; Huang 1999; Kuo 2002; Nayak 2003). However, typical Western diets provide only 1 mg of copper daily, less than even the lower limit of 1.5 to 3.0 mg estimated safe and adequate daily dietary intake (ESADDI) of copper (Kelvay 1998; Failla 1999; Ma 2000; Pang 2001; Davis 2003). Therefore, dietary copper supplementation is likely necessary for disulfiram to be maximally effective as an antineoplastic drug. We project that the optimal dose of copper supplementation to pair with disulfiram is 8 mg elemental copper a day, the upper level of recommended daily copper (Institute for Medicine 2002), administered as copper gluconate, a substance generally regarded as safe (GRAS) (Code of Federal Regulation 2004). This amount would provide an eight-fold higher intake of copper than most American adults consume daily. Large amounts of ingested copper could result in hepatic failure and hemolysis similar to that seen with Wilson's disease, the rare genetic syndrome from hyperabsorption of copper. However, 8 mg of elemental copper has been previously administered to humans with few untoward effects (Pratt 1985; Olivares 1996; Rosado 2003; Mendez 2004; Araya 2005), and in one study even 20 mg of daily copper supplementation was well-tolerated (Araya 2004). Although copper intake is homeostatically regulated, with reduced gastrointestinal absorption at high intakes (Turnland 2005), chronic ingestion of as much as 60 mg elemental copper daily is likely toxic to normal individuals (O'Donohue 1993). In combining copper gluconate with disulfiram as an antineoplastic strategy, we would propose to administer the two in a fashion similar to that used for treatment of our patient with metastatic ocular melanoma, who experienced no diarrhea from zinc gluconate and disulfiram given at different times of the day (Figure 6.10). Copper gluconate containing up to 8 mg elemental copper would be given in the morning a half hour before breakfast, and disulfiram would be consumed with the evening meal. The rationale for separating administration of the two agents in time is to avoid producing gastrointestinal toxicity such as mucositis from complexation of copper by disulfiram in the gut.

Administered separately, we believe that disulfiram and Cu2+ will complex in vivo, forming a bis(diethyldi-thiocarbamato)-copper(II) complex (Johansson 1992) that will provide enhanced antineoplastic activity. It is also possible that metabolites of disulfiram have important activities (Loo 2004) that might also be enhanced by supplementation with copper. Administered orally, both disulfiram and Cu2+ will likely achieve high hepatic concentrations before distribution to other body tissues. This might suggest a utility of disulfiram and Cu2+ in treating primary hepatic tumors such as hepatomas, or secondary hepatic metastases from common malignancies such as colonic adenocarcinoma. The possibility of selective hepatic antineoplastic activity is supported by our experience with the patient suffering from metastatic ocular melanoma (Figure 6.10).

Subjects in this study will include those with advanced cancers metastatic to the liver who are not currently receiving or are eligible for other therapeutic approaches. When prescribed clinically for alcohol aversion, disulfiram is indicated in doses ranging from 125 mg to 500 mg orally each day. For safety reasons, we will initiate disulfiram use at a fixed dose of 250 mg per day, given with the evening meal. We will begin dosing with copper gluconate (2 mg elemental copper) given daily with the morning breakfast meal. These dose times are chosen to separate in time the administration of copper gluconate and disulfiram so that they will not be within the gastrointestinal lumen simultaneously, thereby preventing development of diarrhea and other side effects of mucositis from intraluminal formation of metal-thiocarbamate complexes. Copper gluconate doses will be increased in cohorts of 3 to 6 patients as detailed below as long as dose limiting toxicity is not observed. The maximum dose of copper gluconate to be administered will be the equivalent of 8 mg of elemental copper for the reasons outlined above. Subjects will be maintained on this regimen and followed for the duration of the protocol as long as they are not showing toxicity or disease progression, with periodic measurement of end-points outlined later. Major emphasis will be placed on following ALT and AST as indices of safety and serial abdominal imaging to determine the anatomic burden of hepatic metastases. During the protocol and for four weeks thereafter, subjects will be warned against the ingestion of ethanol and against exposure to alcohol-containing medications or consumer products.

We propose the gradually escalated dosing scheme above in anticipation of the most likely toxicity of the combined ingestion of disulfiram and copper supplements: hepatotoxicity. After gastrointestinal absorption, both agents are likely to be concentrated first in the liver. Therefore, the greatest risk will likely be an increase in hepatic transaminases. From experience with the combined administration of disulfiram and zinc supplements to a patient (Brar 2004) we believe that separating the times at which copper gluconate (morning breakfast meal) and disulfiram (evening meal) are ingested will prevent bothersome diarrhea or other symptoms of mucositis resulting from metal-thiocarbamate complexation within the bowel lumen. We anticipate that careful warning against the ingestion of ethanol-containing beverages or exposure to alcohol-containing consumer products will avert the risk of an inadvertent disulfiram ethanol reaction.

ELIGIBILITY:
Inclusion Criteria:

The subjects must fulfill all the following inclusion criteria to be eligible for participation in the study, unless otherwise specified:

1. Male and female patients with stage IV cancer with metastases demonstrated on abdominal computed tomography (CT) or MRI imaging; patients may have metastatic disease at other sites than the liver, but should have hepatic metastases in order to be eligible for enrollment on this study. Patients are eligible irrespective of the histologic origin of their malignancy but should have exhausted or be unwilling to undergo standard treatment approaches. If a primary histologic diagnosis of malignancy has not been established, hepatic metastases will have to be biopsy proven. Liver disease should be measurable by RECIST criteria.
2. Age of 18 years or more;
3. ECOG performance status of 0 - 2;
4. Patients must have exhausted all standard avenues of therapy for their cancer if such therapy is available, or should be unwilling to undergo such therapy;
5. Not currently receiving other cancer chemotherapy;
6. Not currently participating in another study;
7. Anticipated survival of at least 3 months;
8. Baseline AST and ALT not greater than 2.5 X upper limit of normal;
9. Serum copper within normal limits
10. Serum ceruloplasmin > 17 mg/dL;
11. Able and willing to provide informed consent and to comply with study procedures;
12. Able to ingest oral medications;
13. No known allergy to disulfiram or copper gluconate;
14. Willing to refrain from ingestion of alcoholic beverages while on the study.

Exclusion Criteria:

Potential study subjects who meet any of the following criteria are not eligible for participation in the study:

1. Participation in another clinical trial of a therapeutic drug during the past 30 days;
2. Addiction to alcohol or cocaine;
3. Baseline AST or ALT greater than 2.5 X upper limit of normal;
4. Unable to ingest oral medications;
5. Unable to undergo CT scanning because of inability to lie recumbent in the scanner;
6. Actively receiving cytotoxic cancer chemotherapy agents;
7. Anticipated survival of less than 3 months;
8. Women of child-bearing potential who are not using a commonly accepted effective means of contraception; women of child-bearing potential will have a pregnancy test before enrollment.
9. History of active liver disease, including chronic active hepatitis, viral hepatitis (hepatitis B, C and CMV), cholestatic jaundice from any etiology, toxic hepatitis, or cholestatic hepatitis or jaundice with bilirubin greater than 2.0 X upper limit of normal;
10. History of Wilson's disease or family member with Wilson's disease;
11. History of hemochromatosis or family member with hemochromatosis;
12. History of other iron overload syndrome such as hemochromatosis.
13. Need for warfarin or theophylline, the metabolism of which is likely influenced by disulfiram.
14. Pregnant women and nursing mothers are not allowed to enroll on this study.
15. Patients who are taking medications metabolized by cytochrome P450 2E1, including chlorzoxazone or halothane and its derivatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determine the safety and toxicity profile of co-administration of disulfiram and copper gluconate for the treatment of refractory malignancies that have metastasized to the liver | July 2011

SECONDARY OUTCOMES:
Determine if disulfiram and copper gluconate induce measurable responses for the treatment of hepatic metastases from solid tumors | July 2011
Qualitative assessment of the induction of S-glutathionylation in proteins of circulating leukocytes in patients treated with disulfiram and copper gluconate | July 2011

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Grossmann, MD, PhD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Kelley KC, Grossman KF, Brittain-Blankenship M, Thorne KM, Akerley WL, Terrazas MC, Kosak KM, Boucher KM, Buys SS, McGregor KA, Werner TL, Agarwal N, Weis JR, Sharma S, Ward JH, Kennedy TP, Sborov DW, Shami PJ. A Phase 1 dose-escalation study of disulfiram and copper gluconate in patients with advanced solid tumors involving the liver using S-glutathionylation as a biomarker. BMC Cancer. 2021 May 7;21(1):510. doi: 10.1186/s12885-021-08242-4. PMID 33957901